CLINICAL TRIAL: NCT02386137
Title: Volumetric MR-HIFU Ablation of Uterine Fibroids: Factors Influencing Intraprocedural Thermal Parameters
Brief Title: Factors Influencing Volumetric MR-HIFU Ablation of Uterine Fibroids
Acronym: PERAGUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2014/05
Record Dates: First submitted 2015-02-18; First posted 2015-03-11 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Uterine Fibroid
Keywords: MR-HIFU; HIFU; Fibroid treatment; MR Perfusion; CEUS perfusion; Diffusion weighted imaging; ARFI; Fibroid stiffness
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient (Experimental): Woman aged more than 18 years having one or two symptomatic fibroid with size < 15cm.
  Interventions: Device: Contrast-enhancement ultrasound with Sonovue

INTERVENTIONS:
Device: Contrast-enhancement ultrasound with Sonovue

SUMMARY:
Magnetic resonance (MR)-guided high-intensity focused ultrasound (HIFU) ablation is increasingly being used worldwide to treat symptomatic uterine fibroids because of its excellent therapeutic efficacy in controlling symptoms and its excellent safety record. Despite the benefits, it should be recognized that MR HIFU ablation does not always yield good therapeutic outcomes. High signal intensity on T2-weighted MR images and a high volume transfer constant (or Ktrans) on dynamic contrast material-enhanced MR images are the most well-known risk factors for poor ablation outcomes as measured with the non-perfused volume (NPV) ratio (ie, NPV divided by fibroid volume).

The aim of this study is to assess the influence of fibroid perfusion (evaluated by MRI and contrast enhanced ultrasound), apparent diffusion coefficient (evaluated by MR-diffusion imaging) and fibroid stiffness (evaluated by ARFI) on ablation efficiency during uterine fibroid treatment by MR-HIFU.

DETAILED DESCRIPTION:
Preprocedural predictors of treatment efficacy will be useful for excluding in advance patients who would not benefit from this treatment, thereby contributing to improved overall clinical outcomes. During ablathermy treatment lost of energy depend of tissue perfusion and thermic diffusion while energy laying depend of tissue absorption coefficient. Study these parameters before treatment could bring important information to the treatment difficulty and its efficacy. The investigators will study and compare fibroid perfusion with dynamic contrast-enhanced magnetic resonance imaging and contrast-enhanced ultrasound (CEUS). CEUS will be performed with contrast agent (SONOVUE). Thermic diffusion could be linked with fibroid stiffness. Fibroid stiffness will be quantified with velocity of shear wave measured by acoustic radiation force impulse (ARFI). Tissue absorption coefficient is correlated with the architecture and the cellularity of the tissue so the investigators think that apparent diffusion coefficient (computed with diffusion weighted imaging) could be correlated with ablathermy efficiency and other intra procedural thermal parameters.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Aged more than 18 years
* Not postmenopausal
* Having one or two symptomatic fibroid with size < 15cm.
* Symptoms Severity Score (SSS) score on Uterine Fibroid Symptoms related Quality of Life (UFS-Qol) ≥ 10
* Signed informed consent prior to any study related procedure
* With a medical insurance

Exclusion Criteria:

* Contraindicated to MR examination, SONOVUE and gadolinium contrast injection (pregnancy etc..).
* Presence or suspicious of pelvic malignant tumor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Ablathermy efficiency. | 2 months after inclusion
  necrosis tumor volume / total volume ratio

SECONDARY OUTCOMES:
Thermal parameters | 2 months after inclusion
  Total duration of insonification Maximal temperature peak Cooling rate Efficient thermal dose Necrosis percentage Processing speed (necrosis volume / processing time) Transmitter/fibroma distance
Fibroid signal intensity ratio on T2. | At inclusion and 2 months after inclusion
  Measurements of influence of fibroid signal intensity ratio on T2 on intraprocedural thermal parameters.
Fibroids perfusion data computed with MR perfusion | At inclusion
  Comparison fibroids perfusion data computed with MR perfusion versus contrast-enhanced ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BENARD, MD, Study Chair — University Hospital Bordeaux, France
Locations (1):
- Service d'imagerie médicale, Bordeaux, France